CLINICAL TRIAL: NCT06941454
Title: Investigating the Effect of Smartphone Usage on Balance and Dual Task Performance in University Students
Brief Title: Effect of Smartphone Usage
Status: Not yet recruiting | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Pelin Tiryaki, PhD, University of Yalova
Other Study IDs: 2209-A/123
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: smartphone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Screen time is defined as the time spent on many electronic and technological devices such as laptops, tablets, televisions, game consoles, and smartphones. The largest portion of screen time is made up of smartphones, which are currently used at very high rates. The increase in screen time, which describes the time an individual spends in front of technological devices, can pave the way for various physical problems when not controlled. The most important of these problems caused by excessive screen use due to increased smartphone use is postural disorders. Based on this, the original value of this research is to examine and reveal the effects of smartphone use on balance and dual-task performance. Scientific data can be reached on the negative effects of increased screen use caused by smartphone use.

DETAILED DESCRIPTION:
Screen time is defined as the time spent on many electronic and technological devices such as laptops, tablets, televisions, game consoles, and smartphones. The largest portion of screen time is made up of smartphones, which are currently used at very high rates. The increase in screen time, which describes the time an individual spends in front of technological devices, can pave the way for various physical problems when not controlled. The most important of these problems caused by excessive screen use due to the increase in smartphone usage times is postural disorders. It was planned to examine and reveal the effects of smartphone usage time on balance and dual-task performance. This study was planned as a prospective cross-sectional study. It was planned to evaluate at least 50 participants. The average smartphone usage times of the participants will be recorded. Static and dynamic balance tests (Y Balance Test and Flamingo Test) will be applied and a cognitive task will be added to these tests by including smartphone usage, thus evaluating dual-task performance. The obtained data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30
* Have a smartphone usage period of the last 7 days

Exclusion Criteria:

* Having a severe medical condition
* Having any disease that may affect cognitive level
* Having any disease that may affect balance
* Being pregnant
* Having an orthopedic or neurological surgery within the last year
* Using a mobility assistive device
* Not owning a smartphone

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Smartphone usage time | Baseline
  The average daily smartphone usage time will be calculated by dividing the total smartphone usage time for the last week by 7. The average smartphone usage time will be recorded in minutes.
Y Balance Test | Baseline
  The Y balance test is a time-efficient test that evaluates the dynamic limits of stability and asymmetric balance in three directions (anterior, posteromedial, and posterolateral). The test setup consists of three tape measures with distances in cm on them, one located anteriorly, the other two posterolaterally and posteromedially.
Flamingo Balance Test | Baseline
  During the test, the participant will be asked to stand on the board with his/her foot, lift his/her other foot off the ground, and hold his/her knee with the same hand to maximum flexion. The stopwatch will be started and the measurement will begin when the participant releases the hand of the researcher from whom he/she receives support. The stopwatch will be stopped when the participant releases his/her foot or when any part of his/her body touches the ground.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Serdar CC, Cihan M, Yucel D, Serdar MA. Sample size, power and effect size revisited: simplified and practical approaches in pre-clinical, clinical and laboratory studies. Biochem Med (Zagreb). 2021 Feb 15;31(1):010502. doi: 10.11613/BM.2021.010502. Epub 2020 Dec 15. PMID 33380887
- [Background] Liebherr, M., Schubert, P., Antons, S., Montag, C., & Brand, M. (2020). Smartphones and attention, curse or blessing? - A review on the effects of smartphone usage on attention, inhibition, and working memory. Computers in Human Behavior Reports, 1, 100005. https://doi.org/10.1016/j.chbr.2020.100005
- [Background] Hill MW, Wdowski MM, Rosicka K, Kay AD, Muehlbauer T. Exploring the relationship of static and dynamic balance with muscle mechanical properties of the lower limbs in healthy young adults. Front Physiol. 2023 May 26;14:1168314. doi: 10.3389/fphys.2023.1168314. eCollection 2023. PMID 37304823
- [Background] Fusco A, Giancotti GF, Fuchs PX, Wagner H, da Silva RA, Cortis C. Y balance test: Are we doing it right? J Sci Med Sport. 2020 Feb;23(2):194-199. doi: 10.1016/j.jsams.2019.09.016. Epub 2019 Sep 26. PMID 31601458
- [Background] Adamczewska-Chmiel K, Dudzic K, Chmiela T, Gorzkowska A. Smartphones, the Epidemic of the 21st Century: A Possible Source of Addictions and Neuropsychiatric Consequences. Int J Environ Res Public Health. 2022 Apr 23;19(9):5152. doi: 10.3390/ijerph19095152. PMID 35564547